CLINICAL TRIAL: NCT05225636
Title: Stroke Process in FEmoral Versus Radial Access
Acronym: SFERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR(AG)209/2021
Record Dates: First submitted 2021-08-27; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Ischemic Stroke, Acute
Keywords: Radial access; Femoral access; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Thrombectomy

STUDY DESIGN:
Intervention Model Description: Randomized, prospective clinical trial, under conditions of routine, open-label clinical practice, with the main objective evaluated by an independent investigator who was not blinded to the treatment received. The study will be single-center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial access (Active Comparator): The ischemic stroke treatment will be performed through the radial artery (as first option)
  Interventions: Procedure: thrombectomy
- Femoral access (Active Comparator): The ischemic stroke treatment will be performed through the femoral artery (as first option)
  Interventions: Procedure: thrombectomy

INTERVENTIONS:
Procedure: thrombectomy — Extraction of intracranial thrombus in an acute large vessel occlusion

SUMMARY:
In patients with suspected acute stroke due to large vessel occlusion with indication for endovascular treatment, radial access is just as safe, fast, and effective as femoral access, and it improves the entire stroke treatment process.

DETAILED DESCRIPTION:
Investigators will compare the procedure times, angiographic results as well as the clinical evolution and the patient's experience during their hospital stay and after discharge, depending on the arterial access practiced for mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high suspicion of ischemic stroke due to large cerebral vessel occlusion defined by NIHSS> 10.
* Immediate availability of the entire team responsible for endovascular treatment (Neurologist, Neurointerventional physician, Anesthetist, Nursing, Technicians ...)
* Radial artery diameter ≥2.5 mm
* Presence of femoral pulse or patency by ultrasonography in its defect.
* Previous functional independence (mRS 0-2).

Exclusion Criteria:

* Life expectancy of less than 6 months.
* Intracranial hemorrhage
* Patients with pre-existing neurological or psychiatric pathology that may confuse future evaluations.
* No availability for follow-up after 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-04-28 (Estimated)

PRIMARY OUTCOMES:
No inferiority of radial access in the recanalization rate | Immediate after treatment
  To demonstrate the non-inferiority of radial access with respect to femoral access in the recanalization rate (% mTICI 2b-3 in 3 or fewer passes) obtained in patients with large vessel occlusion treated by mechanical thrombectomy.

SECONDARY OUTCOMES:
No differences in complications in vascular access | 24 hours
  Comparison in frequency of access vessel occlusion, bleeding or presence of pseudoaneurysm
Grades of modified Thrombolysis in Cerebral Infarction | 24 hours
  Grade of recanalization after first pass, third pass and at the end of the procedure
Change of artery access | 24 hours
  Rate of need to change from radial to femoral access and from femoral to radial access
Patient Reported Outcomes | 5 days
  PROMS Patient Reported Outcomes Measures
Patient experience | 5 days
  PREMS Patient Reported Experience Measures
Degree of disability/dependence after a stroke | 24 hours and at 90 days
  modified rankin scale (from 0 to 6, being 0 best and 6 worst)
Times during hospitalization | At 24 hours and during first 5 days
  Beginning of sitting, ambulation, rehabilitation and total time of hospital admission, need for urinary catheter

CONTACTS AND LOCATIONS:
Overall Officials: ALEJANDRO TOMASELLO, MD, Principal Investigator — Hospital Universitari Vall d'Hebron Research Institute
Locations (2):
- Spain (2):
  - Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
After finishing the study we will share all the data if a collaboration is proposed
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publishing our paper
Access Criteria: We will share the data for collaborate with other institutions.

REFERENCES:
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Saver JL, Goyal M, van der Lugt A, Menon BK, Majoie CB, Dippel DW, Campbell BC, Nogueira RG, Demchuk AM, Tomasello A, Cardona P, Devlin TG, Frei DF, du Mesnil de Rochemont R, Berkhemer OA, Jovin TG, Siddiqui AH, van Zwam WH, Davis SM, Castano C, Sapkota BL, Fransen PS, Molina C, van Oostenbrugge RJ, Chamorro A, Lingsma H, Silver FL, Donnan GA, Shuaib A, Brown S, Stouch B, Mitchell PJ, Davalos A, Roos YB, Hill MD; HERMES Collaborators. Time to Treatment With Endovascular Thrombectomy and Outcomes From Ischemic Stroke: A Meta-analysis. JAMA. 2016 Sep 27;316(12):1279-88. doi: 10.1001/jama.2016.13647. PMID 27673305
- [Background] Mazighi M, Chaudhry SA, Ribo M, Khatri P, Skoloudik D, Mokin M, Labreuche J, Meseguer E, Yeatts SD, Siddiqui AH, Broderick J, Molina CA, Qureshi AI, Amarenco P. Impact of onset-to-reperfusion time on stroke mortality: a collaborative pooled analysis. Circulation. 2013 May 14;127(19):1980-5. doi: 10.1161/CIRCULATIONAHA.112.000311. PMID 23671178
- [Background] Jolly SS, Amlani S, Hamon M, Yusuf S, Mehta SR. Radial versus femoral access for coronary angiography or intervention and the impact on major bleeding and ischemic events: a systematic review and meta-analysis of randomized trials. Am Heart J. 2009 Jan;157(1):132-40. doi: 10.1016/j.ahj.2008.08.023. Epub 2008 Nov 1. PMID 19081409
- [Background] Valgimigli M, Gagnor A, Calabro P, Frigoli E, Leonardi S, Zaro T, Rubartelli P, Briguori C, Ando G, Repetto A, Limbruno U, Cortese B, Sganzerla P, Lupi A, Galli M, Colangelo S, Ierna S, Ausiello A, Presbitero P, Sardella G, Varbella F, Esposito G, Santarelli A, Tresoldi S, Nazzaro M, Zingarelli A, de Cesare N, Rigattieri S, Tosi P, Palmieri C, Brugaletta S, Rao SV, Heg D, Rothenbuhler M, Vranckx P, Juni P; MATRIX Investigators. Radial versus femoral access in patients with acute coronary syndromes undergoing invasive management: a randomised multicentre trial. Lancet. 2015 Jun 20;385(9986):2465-76. doi: 10.1016/S0140-6736(15)60292-6. Epub 2015 Mar 16. PMID 25791214
- [Background] Chase AJ, Fretz EB, Warburton WP, Klinke WP, Carere RG, Pi D, Berry B, Hilton JD. Association of the arterial access site at angioplasty with transfusion and mortality: the M.O.R.T.A.L study (Mortality benefit Of Reduced Transfusion after percutaneous coronary intervention via the Arm or Leg). Heart. 2008 Aug;94(8):1019-25. doi: 10.1136/hrt.2007.136390. Epub 2008 Mar 10. PMID 18332059
- [Background] Bertrand OF, Belisle P, Joyal D, Costerousse O, Rao SV, Jolly SS, Meerkin D, Joseph L. Comparison of transradial and femoral approaches for percutaneous coronary interventions: a systematic review and hierarchical Bayesian meta-analysis. Am Heart J. 2012 Apr;163(4):632-48. doi: 10.1016/j.ahj.2012.01.015. PMID 22520530
- [Background] Kolkailah AA, Alreshq RS, Muhammed AM, Zahran ME, Anas El-Wegoud M, Nabhan AF. Transradial versus transfemoral approach for diagnostic coronary angiography and percutaneous coronary intervention in people with coronary artery disease. Cochrane Database Syst Rev. 2018 Apr 18;4(4):CD012318. doi: 10.1002/14651858.CD012318.pub2. PMID 29665617
- [Background] Ghani MR, Busa V, Dardeir A, Marudhai S, Patel M, Abdelmoneim YM, Jan A, Eskander N. Mechanical Thrombectomy in Patients With Acute Ischemic Stroke: A Comparison of Transradial Versus Transfemoral Cerebral Angiography. Cureus. 2020 Oct 12;12(10):e10919. doi: 10.7759/cureus.10919. PMID 33194486
- [Background] Phillips TJ, Crockett MT, Selkirk GD, Kabra R, Chiu AHY, Singh T, Phatouros C, McAuliffe W. Transradial versus transfemoral access for anterior circulation mechanical thrombectomy: analysis of 375 consecutive cases. Stroke Vasc Neurol. 2021 Jun;6(2):207-213. doi: 10.1136/svn-2020-000624. Epub 2020 Nov 16. PMID 33199413
- [Background] Chen SH, Snelling BM, Sur S, Shah SS, McCarthy DJ, Luther E, Yavagal DR, Peterson EC, Starke RM. Transradial versus transfemoral access for anterior circulation mechanical thrombectomy: comparison of technical and clinical outcomes. J Neurointerv Surg. 2019 Sep;11(9):874-878. doi: 10.1136/neurintsurg-2018-014485. Epub 2019 Jan 22. PMID 30670623
- [Background] Khanna O, Mouchtouris N, Sweid A, Chalouhi N, Ghosh R, Al Saiegh F, Gooch MR, Tjoumakaris S, Rosenwasser RH, Romo V, Jabbour P. Transradial approach for acute stroke intervention: technical procedure and clinical outcomes. Stroke Vasc Neurol. 2019 Nov 27;5(1):103-106. doi: 10.1136/svn-2019-000263. eCollection 2020. PMID 32411415
- [Background] Crockett MT, Selkirk GD, Chiu AHY, Singh TP, McAuliffe W, Phillips TJ. First line transradial access for posterior circulation stroke intervention; initial 12-month experience at a high volume thrombectomy center. J Clin Neurosci. 2020 Aug;78:194-197. doi: 10.1016/j.jocn.2020.04.069. Epub 2020 Apr 23. PMID 32336634
- [Background] Maud A, Khatri R, Chaudhry MRA, Vellipuram A, Cruz-Flores S, Rodriguez GJ. Transradial Access Results in Faster Skin Puncture to Reperfusion Time than Transfemoral Access in Posterior Circulation Mechanical Thrombectomy. J Vasc Interv Neurol. 2019 May;10(3):53-57. PMID 31308872
- [Background] Khanna O, Sweid A, Mouchtouris N, Shivashankar K, Xu V, Velagapudi L, Stricsek G, Amllay A, Texakalidis P, Gooch MR, Tjoumakaris S, Rosenwasser RH, Jabbour PM. Radial Artery Catheterization for Neuroendovascular Procedures. Stroke. 2019 Sep;50(9):2587-2590. doi: 10.1161/STROKEAHA.119.025811. Epub 2019 Jul 17. PMID 31311466
- [Background] Amoroso G, Sarti M, Bellucci R, Puma FL, D'Alessandro S, Limbruno U, Canova A, Petronio AS. Clinical and procedural predictors of nurse workload during and after invasive coronary procedures: the potential benefit of a systematic radial access. Eur J Cardiovasc Nurs. 2005 Sep;4(3):234-41. doi: 10.1016/j.ejcnurse.2005.03.005. PMID 15914085
- [Derived] Hernandez D, Requena M, Olive-Gadea M, de Dios M, Gramegna LL, Muchada M, Garcia-Tornel A, Diana F, Rizzo F, Rivera E, Rubiera M, Pinana C, Rodrigo-Gisbert M, Rodriguez-Luna D, Pagola J, Carmona T, Juega J, Rodriguez-Villatoro N, Molina C, Ribo M, Tomasello A. Radial Versus Femoral Access for Mechanical Thrombectomy in Patients With Stroke: A Noninferiority Randomized Clinical Trial. Stroke. 2024 Apr;55(4):840-848. doi: 10.1161/STROKEAHA.124.046360. Epub 2024 Feb 1. PMID 38299334